CLINICAL TRIAL: NCT06869759
Title: Effectiveness of Community Health Workers Induced Prevention of Breast Cancer by Community Health Promotion and Education Implementation Strategies in Jumla - a Cluster Randomised Controlled Trial
Brief Title: "Effectiveness of Community Health Workers in Breast Cancer Prevention in Jumla: a Cluster Randomized Trials
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karnali Academy of Health Sciences (Other)
Responsible Party: Principal Investigator, Bharat Kafle, Fellowship, Karnali Academy of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BC2024
Record Dates: First submitted 2025-01-08; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer; Prevention
Keywords: Health Promotion and Education Strategies
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Arm (Experimental): Arm Description: Clusters will be based on the municipality's wards, to measure the effectiveness of implementation outcomes. There are nine wards in the study site, three of which will be selected for intervention group. Thirty samples will be obtained from each randomly selected cluster of intervention.
  Interventions: Behavioral: Implementation strategy - Health Promotion and Education-based intervention
- Control Arm (No Intervention): Arm Description: Thirty samples will be obtained from each randomly selected cluster of control group who would not be given any intervention, this group consist of 90 participants. The usual work done by the health system of Nepal (i.e: PEN package); after the end line, will also capacitate the control group by radio jingle after seven month of intervention. A mass campaign will be conducted on the process and importance of BSE by airing a radio jingle on local FM.

INTERVENTIONS:
Behavioral: Implementation strategy - Health Promotion and Education-based intervention — Firstly, three broad strategies will be implemented in the intervention arm (use of advisory boards, sensitization, and linkage to care). The advisory board meetings will be held every month to discuss the progress and receive their feedback. Secondly, orientation and capacity building will be done by onsite coaching to community health workers at the health facility level on BSE. Those trained health workers will frequently capacitate FCHVs during monthly meetings. Then, FCHV will visit the community to be aware of BSE as well as they will be involved in a stigma reduction campaign. Sensitization to FCHVs through orientation and capacity building by providing 3 batch training to selected 3 wards, then FCHVs aware and practice the skills of BSE to the recruited participants during home visit and Thirdly, the suspected and identified cases will be linked by strengthening the referral mechanism of the health system and CHWs reminders for follow-up to cases.
  Arms: Intervention Arm

SUMMARY:
Breast cancer is the second most prevalent cancer among Nepali females, accounting for 17.1% of cases and 7.7% of female cancer-related deaths. It is more common in younger, premenopausal women, often diagnosed at advanced stages. Raising awareness through community education is crucial for promoting breast cancer screening, particularly in low-resource settings like Nepal, where clinical breast exams are essential early detection tools. Integrating breast cancer education into the health system can enhance knowledge, encourage screening, and promote healthy behaviors for prevention. Early detection significantly improves treatment outcomes and survival rates.

In remote areas, limited access to advanced detection technologies makes breast self-examination (BSE) the most feasible and cost-effective method, particularly in Jumla. This study evaluates the effectiveness of community health worker-led breast cancer prevention through health promotion and education strategies. It follows PROCTOR's framework and the Health Belief Model (HBM) A mixed-methods design will be employed, incorporating an embedded implementation science approach, a cluster-randomized trial, and mixed-method research. The study population includes married women of Jumla, female community health volunteers (FCHVs), and auxiliary nurse midwives (ANMs). Exclusion criteria include married women ≥20 years old with existing cases of cancer, pregnant or lactating women, FCHVs unable to acquire BSE skills, and untrained ANMs. The sample consists of 90 participants in both intervention and control groups.

Acceptability, Appropriateness, and Feasibility will be assessed using the Acceptability of Intervention Measure (AIM) tool. SOP-based checklists will evaluate fidelity, while FGDs and KIIs will collect qualitative data. Quantitative data will be analyzed using frequency, percentage, mean, and standard deviation. A paired t-test and mixed-effect linear regression will assess effectiveness, while qualitative data will undergo thematic analysis. Findings will be reported per CONSORT guidelines.

Ethical approval will be obtained from the Nepal Health Research Council. Expected outcomes include improved breast cancer knowledge, perception, and screening intention, leading to early detection and reduced prevalence. However, selection bias in cluster trials may limit generalizability.

ELIGIBILITY:
Inclusion Criteria:

* Married women >= 20 years of age group women of CNMP Jumla,
* FCHV, those who can read, write, and understand, and
* ANM

Exclusion Criteria:

* Married women >= 20 years age group women who had a positive existing case,
* Pregnant and lactating women of CNMP Jumla,
* FCHV those who cannot acquire the minimum skill of breast self-examination,
* ANM who untrained for BSE.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — In the quantitative study design, participants will be married women and health facilities. For the qualitative study, the population will be married women of CNMP Jumla. Similarly, community health workers FCHV and CHW will participate in the study.
Enrollment: 180 (Actual)
Dates: Start 2024-08-25 (Actual); Primary Completion 2025-08-25 (Estimated); Study Completion 2025-09-25 (Estimated)

PRIMARY OUTCOMES:
The implementation outcome will be measured by: Acceptability (attitude and perception of women toward BSE and satisfaction levels of the individuals who perform BSE). | From date of randomization, baseline data collection within 2 weeks, and endline 2 months after intervention
  Acceptability (attitude and perception of women toward BSE and satisfaction levels of the individuals who perform BSE). The following indicators will measure this: participants' attitudes toward BSE, perception scores measured in the mean score and SD, and the percentage of women satisfied with BSE practices.
Adoption | From date of randomization, baseline data collection within 2 weeks, and endline 2 months after intervention
  Adoption will be measured by the percentage of CHW and FCHVs willing to adopt BSE. It will also be measured by the extent to which FCHVs are eager and able to integrate BSE activities into their existing roles and responsibilities.
Appropriateness | From date of randomization, baseline data collection within 2 weeks, and endline 2 months after intervention
  Appropriateness will be measured using indicators of the extent to which CNMP is suitably suited to the cultural, social, and economic context and aligned with the needs and preferences of the target population.
Feasibility of implementing FCHV induced breast-self examination | From date of randomization, baseline data collection within 2 weeks, and endline 2 months after intervention
  Feasibility will be measured by assessing the practicality and ease of implementing FCHV in CNMP, quantified through the percentage of health facilities equipped with necessary resources, including training materials and equipment, as well as the proportion of FCHV implementation strategies successfully adopted
Fidelity | From date of randomization, baseline data collection within 2 weeks, and endline 2 months after intervention
  Fidelity will be measured by evaluating the extent to which FCHVs and HFs adhere to the prescribed guidelines and protocols for BSE screening and referral, monitoring the consistency of FCHV discussed in the HMG meeting across different communities, and evaluating the extent to which women adhere to the prescribed guidelines for BSE.
Effectiveness | From date of randomization, baseline data collection within 2 weeks, and endline 2 months after intervention
  Effectiveness outcomes will be measured using the following indicators: Perception, attitude, knowledge, coverage of BSE screening, and Follow-up rates for positive cases.

CONTACTS AND LOCATIONS:
Overall Officials: Bharat Kafle, Principal Investigator — Karnali Academy of Health Sciences
Locations (1):
- Karnali Academy of Health Sciences, Jumla, Karnali, Nepal, Jumla, Karnali, Nepal

IPD SHARING:
Plan to Share IPD: No